CLINICAL TRIAL: NCT01926067
Title: Monitoring of Cardiac Function With 3-axis Accelerometers During Weaning of Cardiopulmonary by Pass After Heart Surgery
Brief Title: Monitoring of Cardiac Function With 3-axis Accelerometers
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2305 A (REK)
Record Dates: First submitted 2012-06-19; First posted 2013-08-20 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Accelerometer; Cardiopulmonary by pass

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim of the study: To validate accelerometers for continuous monitoring of global cardiac function during weaning from cardiopulmonary bypass (CPB) in cardiac surgery.

DETAILED DESCRIPTION:
Hypothesis:

The following hypothesis will be tested: Accelerometer measures are clinical relevant indices of global left and right myocardial performance during weaning from cardiopulmonary bypass.

Model:

The performance of the accelerometer will be tested in a intraoperative setting, during weaning from cardiopulmonary bypass. Accelerometer measures of ventricular systolic and diastolic function will be compared to corresponding measures and indices of ventricular functions by echocardiography and hemodynamic monitoring during a step wise controlled weaning from cardiopulmonary bypass, ensuring precise control of pre- and afterload.

ELIGIBILITY:
The hypothesis will be tested in 20 elective patients.

Inclusion Criteria:

* Significant aortic valvular disease scheduled to undergo cardiac surgery with an estimated extracorporeal circulation time > 40 min.

Exclusion Criteria:

* Evolving myocardial infarction,
* dyskinetic wall motions,
* cardiogenic shock,
* hepatic dysfunction or esophageal disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant aortic stenosis scheduled for surgical AVR
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Comparison of global heart function measures between accelerometer, echocardiography and hemodynamics. | The patients will be followed during surgery, approximately 3 hours.
  Measures will be assessed at baseline before cardiopulmonary by pass, at different workloads during a stepwise weaning, and after the cannulas are removed. The accelerometer measurements will be compared to echocardiography and hemodynamics (stroke volume and cardiac output). Systolic global function will be assessed by comparing peak systolic velocity and displacement by the accelerometer and the corresponding findings in echocardiography. The accelerometer systolic measures will also be correlated to ejection fraction with echocardiography. Diastolic global function early inflow (E'), atrial inflow velocity (A') and E'/A' with accelerometers and echocardiography will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, Professor, Study Director — Oslo University Hospital, The Intervention Sentre
Locations (1):
- Oslo University Hospital, The Intervention Sentre, Oslo, Norway

REFERENCES:
- [Derived] Grymyr OH, Beitnes JO, Eidet J, Tollofsrud S, Fiane A, Skulstad H, Fosse E, Halvorsen PS. Detection of intraoperative myocardial dysfunction by accelerometer during aortic valve replacement. Interact Cardiovasc Thorac Surg. 2017 Feb 1;24(2):188-195. doi: 10.1093/icvts/ivw326. PMID 28364479